CLINICAL TRIAL: NCT00418158
Title: Pulmonary Complications After Heart Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catharina Ziekenhuis Eindhoven (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: poho studie
Record Dates: First submitted 2007-01-03; First posted 2007-01-04 (Estimated); Last update posted 2009-11-10 (Estimated); Status verified 2009-11

CONDITIONS: Heart Surgery
Keywords: Pulmonary complications
MeSH Terms: interventions — Therapeutics

INTERVENTIONS:
Behavioral: use of Airlife (therapy)

SUMMARY:
Abstract: Post-operative pulmonary complications after cardiac surgery

Background The Catharina Hospital performs approximately 1700 heart operation each year. One third of the patients stay at the Catharina hospital during their entire post-operative period. Two years ago they abolished the pulmonary support by a physiotherapist. Subjectively, the pulmonary complications increased over the last two years. During an investigation of the contentment of the patients an increase of the pulmonary problems came forward after eliminating the pulmonary support. There have been no further examinations to the pulmonary complications post-operatively.

Objectives The aim of this study is to give the department of cardio-thoracic surgery an advice about the post-operative pulmonary support for patients who underwent heart surgery.

During the study a budgetary analysis will be made.

Methods 120 patients are prospectively randomised in three groups. Randomisation takes place through block randomisation every three weeks. 40 patients will be supported by a physiotherapist. Another 40 patients will be supported by the nurses on the cardiothoracic surgery ward and the last 40 patients will use an incentive therapy with 'Airlife' by a self-management method.

The study population are all patients undergoing heart surgery and spend their entire post-operative period at the Catharina Hospital. In- and exclusion criteria are specified in the protocol on pages 3 and 4.

Outcome The primary outcome is to qualify the pulmonary complications within the three groups. These complications will be objectified by measuring peak flow, an instrument to determine the lung function, and an x-ray of the thorax.

The secondary outcome is the contentment of the patient, which will be determined by a VAS-score (Visual Analogue Scale).

Risks There are no risks for the patient when participating on this study. The patient will have to fill in the VAS-score and measure lung function with the peak flow at two different moments. The study takes place in a clinical setting. There is no extra insurance in conformity with the advice of the METC.

ELIGIBILITY:
Inclusion Criteria:

* Euroscore < 8
* Age > 18 year
* Patients whereby ECC is peri-operatively used
* No psychological history
* Informed consent obtained
* Follow -up at Catherina Hospital

Exclusion Criteria:

* COPD
* Mitral valve plasty or reconstruction
* Off-pump
* Cognitive problems
* Expected comlpications during operation
* Patients with decompensation
* Day 5 post- ok thoracic drains insitu
* Pain score grater than 4
* Abnormal chest x-ray

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2005-12; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: F.J. ter Woorst, MD, Principal Investigator — Catharina Hospital Eindhoven, department of CardioThoracic Surgery. The Netherlands
Locations (1):
- Catharina Hospital, Eindhoven, Netherlands